CLINICAL TRIAL: NCT04396275
Title: The Effect of Cooked Whole Navy Beans and Yellow Peas on Short-term Satiety and Food Intake in Children
Brief Title: The Effect of Navy Beans and Yellow Peas on Satiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-002
Record Dates: First submitted 2020-04-01; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Food; Eating; Satiety; Physical Comfort
Keywords: Pulses; Satiety; Food intake; Appetite; Beans; Peas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cooked whole navy beans (Experimental): A meal consisting of cooked navy beans
  Interventions: Other: Food-1
- Cooked whole yellow split peas (Experimental): A meal consisting of cooked yellow peas
  Interventions: Other: Food-2
- Cooked rice (control) (Experimental): A meal consisting of cooked rice
  Interventions: Other: Food-3

INTERVENTIONS:
Other: Food-1 — Cooked whole navy beans (300 kcal)
  Arms: Cooked whole navy beans
Other: Food-2 — Cooked whole yellow split peas (300 kcal)
  Arms: Cooked whole yellow split peas
Other: Food-3 — Cooked rice considered as control (300 kcal)
  Arms: Cooked rice (control)

SUMMARY:
The frequent consumption of pulses is associated with multiple cardiometabolic benefits in adults including a lower risk for overweight and obesity. However, it remains unclear whether these effects are mediated through the short-term mechanisms, including enhanced satiety and reduced food intake (FI), or through the long-term metabolic effects triggered by regular consumption of pulses. The objective of this study is to investigate the short-term effect of cooked pulses served in the amount similar to their recommended serving of 175ml (3/4 cup) on food intake in 12-14y children, and gastrointestinal comfort over 2-hours. The secondary objective is to evaluate how children perceive the sensory characteristics of the meals made with the whole pulses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy boys and girls born at full-term
* do not receive any medications

Exclusion Criteria:

* Food sensitivities or allergies
* Dietary restrictions
* Health problems
* Learning, emotional or behavioral problems.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Food intake | 120 min
  The amount of energy (kcal) consumed ad libitum with the breakfast meal or water control and with the test meal (pizza lunch) two hours later.
Subjective appetite | 0-120 min
  The subjective assessment of appetite parameters including desire to eat, fullness, hunger and a prospective food consumption measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., for the hunger scale, 0 mm means not hungry at all, and 100 mm means very hungry).
Subjective feeling of physical comfort | 0-120 min
  The subjective assessment of wellness and gastrointestinal symptoms including a feeling of nausea, diarrhea, flatulence, and other parameters measured with 100 mm Visual Analogue Scales with two opposite statements at each end.

SECONDARY OUTCOMES:
Subjective perception of food palatability (pleasantness) | 0, 120 min
  The pleasantness of the meals measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., 0 mm means that food is not pleasant at all, and 100 mm means that the food is very pleasant).

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No